CLINICAL TRIAL: NCT06474546
Title: The Role of Diet, as Mediated by the Gut Microbiome, on Childhood Arthritis Disease Activity: a Feasibility Intervention Study
Brief Title: Feasibility of a Diet Intervention for Juvenile Arthritis
Acronym: DIGEST-JA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Brian M. Feldman, Division Chief Rheumatology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000080845
Record Dates: First submitted 2024-06-05; First posted 2024-06-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Arthritis, Juvenile; Arthritis, Childhood; Juvenile Idiopathic Arthritis
Keywords: arthritis; diet; microbiome
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Diet (MedDiet)
  Interventions: Other: Diet intervention

INTERVENTIONS:
Other: Diet intervention — A diet based on the principles of the Mediterranean Diet (MedDiet): consists of an abundance of plant foods - unrefined cereals, fruit, vegetables, and extra-virgin olive oil - a moderate consumption of poultry, dairy products, eggs, and low consumption of sweets and red meats.
  All subjects will be instructed to follow the MedDiet for 8 weeks by the study team. Families will be given the option to continue for 12 weeks if they wish to do so.

SUMMARY:
Families of children with arthritis are highly interested in the benefits of diet to improve their child's disease and future health outcomes. Previous research shows that the germs - bacteria and other organisms - that live in the intestines (gut microbiome) are important to how well immune systems work, and that what people eat changes their gut microbiome. The investigators want to study whether a certain diet - based on the principles of the Mediterranean Diet - will improve arthritis for children and whether it was changes in the microbiome that led to improvement.

Fifty-four participants in this study will change their diet for an 8-week period, and will have the option of remaining on the diet for an additional 4 weeks. At three time points during the study (beginning, 8 weeks, and 12 weeks), participants will provide stool and blood samples, will complete questionnaires about diet and other aspects of lifestyle and health, and will complete a disease assessment by a clinician. From collecting all these samples and information, the investigators will be able to determine if the diet was successful in improving disease activity in children with arthritis and if the gut microbiome was changed as well.

This study will help the investigators figure out if a larger, and more definitive, study like this is possible to do in children with arthritis and will help the investigators design a bigger multinational study to confirm how diet affects disease outcomes and the microbiome in children with arthritis. If successful, this research will provide scientific knowledge to help families make their way through this difficult to- navigate topic.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-18 years
* Diagnosis of JIA (excluding systemic JIA, enthesitis-related arthritis, and rheumatoid factor (RF) positive polyarthritis) as per International League of Associations for Rheumatology (ILAR) criteria. (For this feasibility study, there will be no requirement for any particular level of disease activity.)
* Subjects on stable treatment - i.e., any medical treatment with disease-modifying antirheumatic drugs (DMARDs) and/or systemic or intraarticular corticosteroids, has been unchanged for 8 weeks, and is unlikely to change for 12 weeks as judged by the treating physician.
* Willingness to provide stool samples.
* English or French fluency adequate to answer the study questionnaires, and participate in diet instruction, as judged by the enrolling physician.

Exclusion Criteria:

* Documented specific food allergies, celiac disease.
* Co-morbidities that might impact the tolerability of the study diet, e.g., type I diabetes, peptic ulcer disease, etc.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
(Feasibility 1) Participant accrual rate: | 8-12 weeks
  The proportion of all subjects who are approached that enroll and the accrual frequency at each site.
(Feasibility 2) The proportion of subjects who complete all the various measurement steps | 8-12 weeks
  Including return of the fecal samples, gender identification, completion rate of the food diary, etc.
  The proportion of subjects who continue in the 12-week extension will be recorded.
(Feasibility 3) Nutrient intake | 8-12 weeks
  Measured by the participants completing an ecologic momentary assessment (EMA) food diary and the corresponding Prospective Urban Rural Epidemiology (PURE) scores. The PURE score is calculated based on what the subjects entered in their EMA food diary. The score is from 0-6, with a higher score representing a healthier diet.
(Feasibility 4) Adherence to the MedDiet | 8-12 weeks
  Measured by Mediterranean Diet Quality Index in children and adolescents (KIDMED) a questionnaire that measures adherence to the MedDiet scores. The index ranges from 0-12. The values are classified into three levels: > 8 is optimal MedDiet, 4-7 means improvement needed to adjust intake to MedDiet patterns, and ≤ 3 is low diet quality.
(Feasibility 5) Tolerability of diet intervention | 8-12 weeks
  Tolerability will be measured by the Gastrointestinal Symptom Scale for Kids (GISSK), a well-validated and simple questionnaire, designed for use in juvenile idiopathic arthritis (JIA). There are 2 parts to the scale. A visual analog scale (VAS) from 0-100 where the higher score represents the higher severity of gastrointestinal symptoms. And a 8-part questionnaire that ranges from 0-8 where 0 represents no gastrointestinal symptoms.
(Mediator 1) Changes in the microbiome | 8-12 weeks
  Measured by intestinal microbial ⍺-diversity (a measure representing the number of microbial groups and how evenly balanced they are within the gut), the individual species and functions of gut organisms (through shotgun metagenomics), and short chain fatty acids (SCFAs).
(Mediator 2) Changes in juvenile arthritis disease activity score | 8-12 weeks
  Measured by the Juvenile Arthritis Disease Activity Scale (cJADAS10). This includes the 1) physician's global assessment of disease activity measured on a 10cm visual analog scale (VAS), (2) parent/patient's global assessment of well-being measured on a 10cm VAS, (3) count of joints with active disease up to 10 active joints. The total score ranges from 0-30 with higher number representing a higher juvenile arthritis disease activity score.
(Mediator 3) Changes in functional status | 8-12 weeks
  Measured by the Childhood Health Assessment Questionnaire (CHAQ) (self/parent report scale that is widely used to measure functional status in children with arthritis). The score ranges from 0-3, with a 0 representing no functional disability and 3 representing severe disability.
(Mediator 4) Changes in quality of life | 8-12 weeks
  Measured by the Quality of My Life (QoML) questionnaire (a validated questionnaire to measure well-being). QoML consists of 3 visual analog scales each scored out of 10. Higher scores indicate better quality of life.
(Mediator 5) Changes in gut inflammation | 8-12 weeks
  Measured by fecal calprotectin.
(Mediator 6) Changes in systemic inflammation | 8-12 weeks
  Measured by a blood biomarker panel, a composite measure of immune activation comprising 49 analytes:
  (sCD40L, EGF, Eotaxin, FGF-2, Flt-3 ligand, Fractalkine, G-CSF, GM-CSF, GROα, IFNα2, IFNγ, IL-1α, IL-1β, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p40), IL-12 (p70), IL-13, IL-15, IL-17A, IL-17E/IL-25, IL-17F, IL-18, IL-22, IL-27, IP-10, MCP-1, MCP-3, M-CSF, MDC (CCL22), MIG, MIP-1α, MIP-1β, PDGF-AA, PDGF-AB/BB, RANTES, TGFα, TNFα, TNFβ, VEGF-A, YKL40)

SECONDARY OUTCOMES:
(Confounder 1) Sleep quality | 8-12 weeks
  Measured by FitBit accelerometry
(Confounder 2) Patient-reported Sleep Quality | 8-12 weeks
  Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbances questionnaire. The total score ranges from 0-40 with a higher score representing a poor sleep quality.
(Confounder 3) Physical activity | 8-12 weeks
  Measured by the Godin-Shephard Leisure-Time Physical Activity Questionnaire (GODIN) exercise questionnaire. A total score of 24 or more is active, 14 - 23 is moderately active, and less than 14 units is sedentary.
(Confounder 4) Sex | 8-12 weeks
  Results will be stratified by sex at birth.
(Confounder 5) Gender | 8-12 weeks
  Gender will be collected using the Perceived Similarity to Gender Groups Measure for children and youth.
(Confounder 6) Medication use | 8-12 weeks
  Will be abstracted from the patient chart. Results will be stratified by medication use.
(Confounder 7) Age | 8-12 weeks
  Stratify data by age group (8 - 12 and 13 - 18)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M. Feldman, Principal Investigator — The Hospital for Sick Children
Locations (7):
- Canada (7):
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan